CLINICAL TRIAL: NCT06398418
Title: A Single and Repeat Dosing and Expansion Study of the Safety, Drug Exposure and Clinical Activity of R-5780 in Combination With a PD-1 (Checkpoint Protein on Immune Cells Called T Cells) Pathway Checkpoint Inhibitor in Patients With Solid Tumors
Brief Title: R-5780-01 In Combination With PD-1 Checkpoint Inhibitors (Checkpoint Protein on Immune Cells Called T Cells) in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rise Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RISE R-5780-01
Record Dates: First submitted 2024-04-29; First posted 2024-05-03 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor, Adult; Solid Tumor; Melanoma; Basal Cell Cancer; Squamous Cell Cancer; Adenoma
Keywords: Solid Tumors
MeSH Terms: conditions — Melanoma; Neoplasms, Basal Cell; Neoplasms, Squamous Cell; Adenoma

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Other): R-5780 Probiotic
  Interventions: Drug: R-5780

INTERVENTIONS:
Drug: R-5780 — Probiotic

SUMMARY:
The goal of this study is determine the safety and tolerability of orally taken probiotic (R-5780) in patients currently on a PD-1 Pathway Checkpoint Inhibitor (checkpoint protein on immune cells called T cells) with Solid Tumors.

DETAILED DESCRIPTION:
Patients will take an oral dosage of probiotic (R-5780 and provide patient reported overall feeling and physician scored measure of their tumors. Blood and fecal evaluations of inflammation and assessment of probiotic (R-5780) on fecal levels will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age to 80
* Ability to provide written informed consent
* Unresectable stage III or stage IV melanoma, basal cell carcinoma, or squamous cell carcinoma as per the American Joint Committee on Cancer 2017 Guidelines (8th Edition) regardless of BRAF mutation status and other solid tumors.
* Refractory to anti-PD (checkpoint Protein on Immune Cells called T cells)-1/L1 therapy per RECIST v1.1 defined as subject who has disease progression after receiving at least two complete cycles of ICI (immune checkpoint inhibitors) therapy or disease progression 6 months from initiation of ICI (immune checkpoint inhibitors) therapy while still on active therapy.
* Life expectancy of greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Subjects must have evaluable disease by CT (computer tomography) or MRI (magnet resonance imaging) per RECIST 1.1 criteria or clinically apparent disease that the investigator can follow for response.

Exclusion Criteria:

* Any serious medical condition or laboratory abnormality or psychiatric condition or any other significant or unstable concurrent medical illness (in the opinion of the Investigator) would preclude protocol adherence or would make the safety of the study drug difficult to assess
* Treatment with systemic broad-spectrum antibiotics.
* No active viral infections.
* Coexisting severe chronic diseases other than cancer (autoimmunity, inflammatory diseases)
* Secondary gastrointestinal motility disorders
* History of solid organ transplant or bone marrow transplant
* Prior CAR-T (chimeric antigen receptor) or allogeneic cellular therapy
* Ongoing systemic immunosuppressive therapy, with the exclusion of prednisone (10 mg/day)
* Concurrent therapy with any other investigational agent, vaccine, or device
* Pregnant or breastfeeding or planning to conceive or father a child during the trial period
* Subjects with untreated brain metastasis. Treated brain metastasis are permitted if stable
* More than 4 prior systemic therapies
* Other cancer medications during treatment period are not permitted
* Enrollment in other clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events and their relationship to R-5780 (probiotic) administration | Baseline through Week 4
  To assess the number of participants with treatment-related adverse events after taking R-5780 (probiotic)

SECONDARY OUTCOMES:
Scale (QOLS) | Baseline through End of Study Day 112
  Collect how the patient is feeling on each study visit on the Quality of Life Scale of 30 questions. The Quality of Life scores are summed so that a higher score indicates higher quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Sarah Cannon Research Institute, Nashville, Tennessee, United States